CLINICAL TRIAL: NCT00620230
Title: A Phase I Study to Assess the Safety, Tolerability, Pharmacokinetic Profile and Pharmacodynamic Effect of Single and Multiple Doses of VAK694 in Healthy and Atopic Subjects
Brief Title: Safety and Tolerability of Single and Multiple Doses of VAK694 in Healthy and Atopic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CVAK694A2102
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis, anti-interleukin 4
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: NVP-VAK694
- 2 (Placebo Comparator)
  Interventions: Drug: NVP-VAK694

INTERVENTIONS:
Drug: NVP-VAK694
  Arms: 1
Drug: NVP-VAK694
  Arms: 2

SUMMARY:
This study will evaluate the safety and tolerability of single and multiple doses of VAK694 in healthy volunteers and otherwise healthy volunteers with a history of allergies.

ELIGIBILITY:
Inclusion Criteria:

* History of allergic rhinitis (Part 2 only)

Exclusion Criteria:

* Very low or high body weight
* Heavy or recent smoker
* Exposure to human monoclonal antibodies

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Routine safety observations and pharmacokinetic measurements | throughout the study

SECONDARY OUTCOMES:
Routine safety observations and pharmacokinetic measurements | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (1):
- Novartis Investigator Site, North Miami Beach, Florida, United States